CLINICAL TRIAL: NCT03646838
Title: Family Experiences After International Adoption
Acronym: VF-ADIN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Other Study IDs: D17-P16
Record Dates: First submitted 2018-03-20; First posted 2018-08-24 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Discrimination, Racial
Keywords: International adoption; Family experiences; Adolescents; France
MeSH Terms: conditions — Racism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the types of experiences faced by families in France who have adopted a child internationally. In addition, internationally adopted adolescents are invited to respond to questions about their own personal experiences.

DETAILED DESCRIPTION:
Microaggressions, or "unintended discrimination" related to adoption have been widely investigated in the USA. These microaggressions may relate to both adoptive status and country of origin, or both. However, the prevalence and qualitative characteristics of these events have been seldom studied in other countries. Differences in cultural norms and practices among countries might influence the type and frequency of microaggressions experienced by adopted children and their families. Brief anonymous questionnaires devised to elicit personal experiences related to microaggressions will be distributed by 4 clinical services serving this population (3 pediatric, 1 child psychiatric) and by 2 large adoptive family support networks to adoptive parents in France. Frequencies and relations between experience of micro-aggressions and other variables will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

Parents :

1. Parents of an internationally adopted child, whose placement occurred at least 6 months ago
2. Willing and able to complete a questionnaire

Adolescents :

1. Internationally adopted adolescents who were placed at least 6 months ago
2. Willing and able to complete a questionnaire

Exclusion Criteria:

Parents :

1. Unwilling or unable to complete the questionnaire

Adolescents :

1. Parents are unwilling for child to participate
2. Child is unwilling to participate
3. Unable to understand the questions

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adoptive parents, regardless of the age of their children, as well as adolescents who have been adopted internationally, directly.
Sampling Method: Non-Probability Sample
Enrollment: 991 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Number and type of micro-aggressions experienced by French families who have adopted internationally | parents respond to a questionnaire at a single time point, regarding their experience. Participation is hence limited to the 30 minutes required to complete the questionnaire.
  Parents will respond to a questionnaire regarding their experiences of micro-aggressions as an adoptive family in France, enumerating the types of discrimination (if any) they have encountered, in what context or environment this occurred, and their feelings in response to these experiences. The types of micro-aggressions could include hearing derogatory comments about adoption in general, their child's country of origin or appearance, etc. Parents may also experience well-meaning but uninformed comments ("how much did she cost?") which are also experienced as micro-aggressions. Simple frequency statistics enumerating these experiences will be compiled. These will be compared to basic demographic indicators such as the country of origin of the child, the child's age at adoption, the child's current age, the time interval since adoption, etc.

SECONDARY OUTCOMES:
Number and type of micro-aggressions experienced by internationally adopted adolescents in France | Adolescents respond to a questionnaire at a single time point, regarding their experiences as an adopted person in France. Participation is hence limited to the 30 minutes required to complete the questionnaire.
  Adolescents will respond to a questionnaire regarding their experiences of micro-aggressions as adopted individuals in France, enumerating the types of discrimination (if any) they have encountered, in what context or environment this occurred, and their feelings in response to these experiences. The types of micro-aggressions could include hearing derogatory comments about adoption in general, their country of origin or appearance, etc. Adolescents may also experience well-meaning but uninformed comments ("why did your real parents abandon you?") which are also experienced as micro-aggressions. Simple frequency statistics enumerating these experiences will be compiled. These will be compared to basic demographic indicators such as their country of origin, their age at adoption, their current age, the time interval since adoption, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Odile MD PEROUSE DE MONTCLOS, Principal Investigator — Hospital SAINTE ANNE
Locations (4):
- France (4):
  - Hospital Enfants CHU du BOCAGE, Dijon
  - Hospital SAINTE ANNE, Paris
  - Hospital NECKER, Paris
  - Hospital MIGNOT, Versailles

REFERENCES:
- [Background] Frable DE, Wortman C, Joseph J. Predicting self-esteem, well-being, and distress in a cohort of gay men: the importance of cultural stigma, personal visibility, community networks, and positive identity. J Pers. 1997 Sep;65(3):599-624. doi: 10.1111/j.1467-6494.1997.tb00328.x. PMID 9327589
- [Background] Sue DW, Capodilupo CM, Torino GC, Bucceri JM, Holder AM, Nadal KL, Esquilin M. Racial microaggressions in everyday life: implications for clinical practice. Am Psychol. 2007 May-Jun;62(4):271-86. doi: 10.1037/0003-066X.62.4.271. PMID 17516773